CLINICAL TRIAL: NCT05496595
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation, and Dose Expansion Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of DCBY02 as a Monotherapy in Patients With Advanced or Metastatic Solid Tumors
Brief Title: DCBY02 as a Monotherapy in Patients With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Review of Data, and our other compound is a better option
Sponsor: DynamiCure Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCBY02-101
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Dose escalation to investigate safety, tolerability, and determine recommended phase 2 dose (RP2D) for DCBY02.
  Interventions: Drug: DCBY02
- Part 2: Dose Expansion (Experimental): Dose expansion to further investigate safety, tolerability, and preliminary evidence of antitumor activity and characterize PK and PD of DCBY02.
  Interventions: Drug: DCBY02

INTERVENTIONS:
Drug: DCBY02 — A monoclonal antibody that binds to CD93, DCBY02 will be administered as a single intravenous (IV) infusion on Day 1 in each 21-day cycle.

SUMMARY:
Study DCBY02-101 is a multicenter, open-label, Phase 1 study to assess the effects of anti-CD93 mAb (DCBY02) as a monotherapy in patients with advanced or metastatic solid tumors.

ELIGIBILITY:
Selected Inclusion Criteria:

Male or female patients ≥ 18 years of age.

Histologically or cytologically confirmed incurable or metastatic solid tumors - colorectal, gastric, non-small cell lung, renal cell, breast, hepatocellular, ovarian, cervical cancer, GBM or with a potential benefit from PD-1/PD-L1 blockade where hypoxia is associated with resistance to PD-1 blockade eg, as reported for or head and neck cancer and is not amenable to curative treatment.

The malignancy must have progressed after at least 1 available standard therapy for incurable disease, and the patient has failed or is intolerant to all available therapies known to be active for the malignancy and have meaningful impact on the disease.

Male or female patients ≥18 years of age 2. Histologically or cytologically confirmed incurable or metastatic solid tumors (including but not limited to colorectal, gastric, non-small cell lung, renal cell, breast, hepatocellular, ovarian, cervical, or head and neck cancer; or GBM). The malignancy must have progressed after at least 1 available standard therapy for incurable disease, and the patient has failed or is intolerant to all available therapies known to be active for the malignancy and have a meaningful impact on the disease. The Investigator needs to discuss any available standard options with the patient and document the benefits and risks of all options along with the rationale for recommending the study.

Note: For patients who are intolerant to or refuse standard of care therapy for recurrent disease, reasons must be documented.

3. Patients with unresectable or metastatic solid tumors, except for patients with GBM, must have a lesion that can be biopsied with acceptable clinical risk and agree to have a fresh biopsy at Screening and an on-treatment biopsy. Every effort must be made to take the second biopsy from the same lesion of the biopsy at Screening.

1. A lesion in a previously irradiated area could be biopsied as long as there is objective evidence of progression of the lesion before study enrollment.
2. Starting in Cohort 3, patients must have at least 1 RECIST measurable lesion for inclusion that will not undergo biopsy.

   4. Patients with solid tumors must have at least 1 measurable lesion according to RECIST 1.1 (non-nodal lesions must be ≥ 1.0 cm in the long axis or ≥ double the slice thickness in the long axis; nodal lesions must be ≥ 1.5 cm in the short axis).

a) A lesion in a previously irradiated area is eligible to be considered as a measurable disease as long as there is objective evidence of progression of the lesion before study enrollment.

b) In Cohort 1 and Cohort 2, patients without measurable lesions are eligible. c) Patients with GBM must meet the RANO criteria of measurable disease (10 mm × 10 mm) for the post-gadolinium primary tumor weighted images (T1WI) 5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2. 6. Adequate organ function and bone marrow reserve as indicated by the following laboratory assessments performed within 14 days prior to the first dose of study drug:

1. Bone marrow function: absolute neutrophil count (ANC) ≥ 1500/μL; hemoglobin ≥ 9 g/dL; platelet count ≥ 75,000/μL.
2. Hepatic function: Total serum bilirubin ≤ 1.5 times the upper limit of normal (ULN); serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT), ≤ 3× ULN (≤ 5 × ULN in the presence of hepatic metastases).

Note: Patients with inherited disorders of bilirubin metabolism should be discussed with the Sponsor.

c) Renal function: Creatinine clearance ≥ 30 mL/minute based on Cockcroft-Gault estimation.

d) Coagulation profile: Prothrombin time (PT) - international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Patients on a stable, maintenance regimen of anticoagulant therapy for at least 30 days prior to the first dose of study drug may have PT/INR measurements > 1.5 × ULN if, in the opinion of the Investigator, the patient is suitable for the study. An adequate rationale must be provided to the Sponsor prior to enrollment.

7. Recovered to Grade 1 or baseline from all toxicity associated with previous therapy or have the toxicity established as sequela.

Note: Neuropathy and/or hearing impairment Grade ≤2, any grade alopecia, or autoimmune endocrinopathies with stable replacement therapy are permitted.

8. Female patients of childbearing potential must:

1. Have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at Screening.
2. Agree to use highly effective contraception from the time that the patient provides informed consent until at least 5 months after the last dose of DCBY02.

Examples of highly effective contraception include the following:

i) Combined hormonal contraceptives (containing both estrogen and progesterone) associated with inhibition of ovulation; may be oral, intravaginal, or transdermal) ii) Intra-uterine device iii) Intra-uterine, hormone-releasing system iv) Bilateral tubal occlusion v) Vasectomized partner vi) Sexual abstinence. 9. Male patients who are not surgically sterile must: Agree to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agree to refrain from donating sperm, as defined below:

a) With a female partner of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year and must refrain from donating sperm during the treatment period and for at least 60 days after the final dose of DCBY02.

b) With pregnant female partners, men must remain abstinent or use a condom to avoid exposing the embryo during the treatment period and for at least 60 days after the final dose of DCBY02.

10. Capable of understanding and complying with the protocol and has signed the required informed consent form (ICF). The appropriate ICF must be signed before relevant study procedures are performed. If applicable, the female partner of a male patient understands and signs the pregnant partner's ICF.

Selection Exclusion Criteria 1. Received treatment with systemic anticancer treatments or investigational products within 14 days before the first dose of study drug or 5 half-lives, whichever is shorter.

Note: Low-dose steroids (oral prednisone or equivalent ≤10 mg per day), hormonal therapy for prostate cancer or breast cancer (as adjuvant treatment), and treatment with bisphosphonates and receptor activator of nuclear factor kappa-Β ligand (RANKL) inhibitors are allowed.

Patients with second malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the patient is not on active anticancer therapy. These patients must be discussed with the medical monitor prior to enrollment.

3. Patients with known active central nervous system (CNS) metastases. Patients with previously treated brain metastases may participate provided that:

1. They are stable (i.e., without evidence of progression by magnetic resonance imaging [MRI]) for ≥ 4 weeks prior to the first dose of study drug),
2. All neurologic symptoms have returned to Baseline, and
3. They have no evidence of new or enlarging brain metastases.
4. If signs or symptoms suggest CNS metastases, a brain MRI or CT scan must be performed to confirm the absence of detectable CNS disease within 2 weeks prior to the first dose of study drug.

   Note: The above criteria are not applicable to GBM patients. For GBM, patients may participate if they are on corticosteroids or on stable or decreasing corticosteroid levels exceeding 2 mg/day dexamethasone (or equivalent doses of other steroids) during the last 3 days prior to enrollment, expectation that the patient will need corticosteroid doses > 2 mg/dexamethasone/day or equivalent during the next 3 months.

   4. New York Heart Association Class III or IV heart disease, active ischemia, or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension, or congestive heart failure within the last 3 months.

   5. Patients with systemic arterial thrombotic or embolic events, such as cerebrovascular accident (including ischemic attacks) or hemoptysis within 3 months prior to the first dose of study drug.

   6. Patients with systemic venous thrombotic events (e.g., deep vein thrombosis) or pulmonary arterial events (e.g., pulmonary embolism) within 1 month prior to the start of study drug.

   7. Left ventricular ejection fraction (LVEF) < 50% or below the lower limit for normal institutional level.

   8. Major surgery within 4 weeks and minor surgery within 2 weeks of the first dose of study drug; following surgeries, all surgical wounds must be healed and free of infection or dehiscence.

   9. Patients with marked proteinuria ≥ 2 g/24 hours and/or nephrotic syndrome. Patients with proteinuria 2+ or greater urine dipstick reading should undergo further assessment, e.g., a 24-hour urine collection.

   10. Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, or any other condition, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.

   11. Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections; patients with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Patient has known positive human immunodeficiency virus (HIV) antibody results or acquired immunodeficiency syndrome (AIDS)-related illness; patients with CD4+ T- cell counts ≥ 350 cells/μL and have not had an AIDS-related illness within the past 12 months will be permitted.

   12. Patient is pregnant or lactating. 13. Known allergy or hypersensitivity to any component of the study drug. 14. Known contra-indications to CNS MRI in patients with GBM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs occurring in the first 28 days following DCBY02 administration | 2 years
Frequency and severity of treatment-emergent adverse events (TEAEs) | From first dose to Cycle 2 Day 8 (28 days)

SECONDARY OUTCOMES:
Objective response rate (ORR) as determined per Investigator assessment | 1 year
Duration of response (DOR) as determined per Investigator assessment | 1 year
Disease control rate (DCR) as determined per Investigator assessment | 1 year
Progression free survival (PFS) as determined per Investigator assessment | 1 year
Overall survival (OS) | 1 year
Pharmacokinetic parameters of DCBY02: maximum observed concentration (Cmax) | 2 years
Pharmacokinetic parameters of DCBY02: area under the concentration-time curve (AUC) | 2 years
Pharmacokinetic parameters of DCBY02: clearance (CL) | 2 years
Pharmacokinetic parameters of DCBY02: volume of distribution (Vz) | 2 years
Pharmacokinetic parameters of DCBY02: half-life (t1/2) | 2 years
Parts 1A/2A: Incidence of anti-drug antibody (ADA) and neutralizing antibodies (NAbs) against DCBY02 | 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Honor Health, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No